CLINICAL TRIAL: NCT06477445
Title: Effect of Visual Feedback Balance Training System Combined with Repetitive Facilitative Exercise on Fall Risk After Stroke: a Randomized Control Trial
Brief Title: Visual Feedback Balance Training System Combined with RFE in Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Mingzhou Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Jingzhi Zhang, therapist-in-charge, Nanjing Mingzhou Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NJKF202406002
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combination group (Experimental): Visual feedback balance training system combined with RFE
  Interventions: Device: Visual feedback balance training system; Other: repetitive facilitative exercise
- RFE group (Active Comparator): Repetitive facilitative exercise (RFE)
  Interventions: Other: repetitive facilitative exercise
- CT group (Active Comparator): Conventional therapy (CT)
  Interventions: Other: conventional therapy

INTERVENTIONS:
Device: Visual feedback balance training system — Using an visual feedback balance training system to provide a dynamic balance training platform for patients to perform balance training based on visual feedback.
  Arms: Combination group
Other: repetitive facilitative exercise — Repetitive facilitative exercise (RFE) is a new technology that combines multiple sensory stimuli and achieves facilitation and reinforcement of the reconstruction of paralyzed neural pathways through repeated and extensive directional exercise.
  Arms: Combination group; RFE group
Other: conventional therapy — Basic training, including passive joint movement and activities of daily living exercise.
  Arms: CT group

SUMMARY:
The goal of this clinical trial is to learn if visual feedback balance training system combined with repetitive facilitative exercise (RFE) work to treat stroke in adults. The main questions it aims to answer are:

Does visual feedback balance training system combined with RFE reduce the fall risk of participants? Can the combination of intelligent rehabilitation robot training system and RFE achieve better effects?

Researchers will compare 3 groups (RFE, visual feedback balance training system under RFE, and conventional therapy) to see if visual feedback balance training system and RFE works to treat stroke.

Participants will:

Receive treatment for 4 weeks Receive scale and instrument testing before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* patients (18 to 74 years old) who suffered a first or second unilateral stroke
* chronic stroke (over 6 months from the onset)
* moderate or higher risk of falls (TUG > 15s, or 10-MWT ≤ 0.8m/s)
* ability to understand and follow simple directions

Exclusion Criteria:

* pregnant or lactating
* lower extremity contracture, pain, or trauma
* perceptual, apraxic, or cognitive deficits that lead to inability to follow verbal instructions
* unable to maintain standing posture
* cerebellar lesion
* clinically unstable medical disorders
* inability to provide informed consent

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
time up and go test (TUG) | From enrollment to the end of treatment at 4 weeks
10-meter walk test (10-MWT) | From enrollment to the end of treatment at 4 weeks
Center of gravity loss index | From enrollment to the end of treatment at 4 weeks
  Use the Libra parameters evaluation system included with visual feedback balance training system
Deviation of bilateral center of gravity movement area | From enrollment to the end of treatment at 4 weeks
  Use the Libra parameters evaluation system included with visual feedback balance training system

SECONDARY OUTCOMES:
functional ambulation category scale (FAC) | From enrollment to the end of treatment at 4 weeks
Fugl-Meyer Assessment (FMA) | From enrollment to the end of treatment at 4 weeks
Berg balance scale (BBS) | From enrollment to the end of treatment at 4 weeks